CLINICAL TRIAL: NCT04088604
Title: PhaseⅠStudy of Irinotecan Hydrochloride Liposome Injection (LY01610) About the Safety, Tolerability, Pharmacokinetics (PK)and Preliminary Efficacy in Patients With Advanced Solid Tumors
Brief Title: Irinotecan Hydrochloride Liposome Injection (LY01610) For Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01610/CT-CHN-101
Record Dates: First submitted 2019-08-22; First posted 2019-09-13 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor
Keywords: LY01610; 5-Fu; Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Parallel
Masking Description: None，Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LY01610-Dose Escalation (Experimental): The starting dose was 30 mg/m2 IV and the subsequent dose was increased according to the protocol of 60 mg/m2, 90 mg/m2, 120 mg/m2, 150 mg/m2, 180mg/m2. The interval between the first dose and the second dose was 3 weeks, followed by 2 weeks.
  Interventions: Drug: LY01610 ( Irinotecan hydrochloride liposome injection )
- LY01610-Dose Extension (Experimental): According to the subjects' tolerance, appropriate dose will be selected and the safety, PK characteristics and initial efficacy of LY01610 were further evaluated in 6 - 8 patients. The interval between the first dose and the second dose was 3 weeks, followed by 2 weeks.
  Interventions: Drug: LY01610 ( Irinotecan hydrochloride liposome injection )
- LY01610 with 5-Fu -Dose Escalation (Experimental): Dose Escalation:
  Based on the results of the first stage, three doses of low, medium and high doses were selected in combination with a fixed dose of 5-Fu to determine the DLT, MTD, PK characteristics and the preliminary efficacy. 5-Fu, 400mg/m2 will be administered intravenously on days 1, followed by 600 mg/m2 given as a 22-hour continuous infusion on day 1 and 2, every 2 weeks.
  Interventions: Drug: LY01610 ( Irinotecan hydrochloride liposome injection ) with 5-Fu（Fluorouracil Injection）
- LY01610 with 5-Fu -Dose Extension (Experimental): Similarly, according to the subjects' tolerance, appropriate dose will be selected and the safety, PK characteristics and initial efficacy of LY01610 combined with a fixed dose of 5-Fu were further evaluated in additional 6 - 8 patients.
  In dose escalation and dose extension stages, both LY01610 and fixed dose 5-Fu will be given once every 2 weeks.
  Interventions: Drug: LY01610 ( Irinotecan hydrochloride liposome injection ) with 5-Fu（Fluorouracil Injection）
- Hydrochloride Injection- pharmacokinetics comparative study (Active Comparator): After receiving the MTD of LY01610, another 8 subjects were enrolled and given Irinotecan Hydrochloride Injection（captol ®） (180mg/m2) once every 2 weeks. Upon completion of the pharmacokinetics study, the sponsor will continue to provide the study drug treatment free of charge, and the researcher will conduct treatment and examination according to the subject's situation, without collecting any safety and efficacy data of the subject.
  Interventions: Drug: Irinotecan Hydrochloride Injection（CAMPTO®）

INTERVENTIONS:
Drug: LY01610 ( Irinotecan hydrochloride liposome injection ) — Part1-Dose Escalation and Part1-Dose Extension : subjects take LY01610;
  Arms: LY01610-Dose Escalation; LY01610-Dose Extension
Drug: LY01610 ( Irinotecan hydrochloride liposome injection ) with 5-Fu（Fluorouracil Injection） — Part2-Dose Escalation and Part2-Dose Extension : subjects take LY01610 with 5-Fu;
  Arms: LY01610 with 5-Fu -Dose Escalation; LY01610 with 5-Fu -Dose Extension
Drug: Irinotecan Hydrochloride Injection（CAMPTO®） — Irinotecan Hydrochloride Injection（CAMPTO®） pharmacokinetics comparative study
  Arms: Hydrochloride Injection- pharmacokinetics comparative study

SUMMARY:
This is a Phase I, open-label, non-randomized, dose-escalation study to evaluate the safety and tolerability, the maximum tolerated dose (MTD) and the dose limited toxicity(DLT) of LY01610 monotherapy and combine with 5-Fu in patients with advanced solid tumors. Additionally, the pharmacokinetics and preliminary efficacy of LY01610 monotherapy and combine with 5-Fu will be investigated in this study.

DETAILED DESCRIPTION:
This study will be conducted in two stages: In the first stage, ascending doses of LY01610 will be administered as monotherapy in participants with solid tumors. The starting dose was 30 mg/m2 and the subsequent dose was increased according to the protocol of 60 mg/m2, 90 mg/m2, 120 mg/m2, 150 mg/m2, 180mg/m2. Each subject received only one dose of the drug, and the next dose group study could only be performed if the previous dose group was completed 21 days of observation after the first dose and safe tolerance was confirmed. According to the subjects' tolerance, appropriate doses will be selected and the safety, PK characteristics and initial efficacy of LY01610 were further evaluated in additional 6 - 8 patients. The interval between the first dose and the second dose was 3 weeks, followed by 2 weeks.Another 8 subjects were enrolled and given CAMPTO® (180 mg/m2) once every 2 weeks to perform the pharmacokinetic profiles.

The second stage is a dose escalation study of LY01610 combined with 5-Fu. Based on the results of the first stage, three doses of low, medium and high doses were selected in combination with a fixed dose of 5-Fu to determine the DLT and MTD. Similarly, according to the subjects' tolerance, appropriate dose will be selected and the safety, PK characteristics and initial efficacy of LY01610 combined with a fixed dose of 5-Fu were further evaluated in 6 - 8 patients. The drug was administered every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 70 years (18 years and 70 years are inclusive).
* Histologically or cytologically confirmed solid tumor for which failed or could not •tolerate standard treatment, or standard effective treatment does not exist.
* The patient should have at least one measurable lesion as the target lesion (according to RECIST 1.1 criteria).
* The predictable survival duration ≥ 3 months.
* The Eastern Cooperative Oncology Group (ECOG) performance status score < 2 point.
* Laboratory results during screening:
* Hematology: Absolute neutrophil count ≥ 1.5× 109/L, platelet count≥ 100× 109/L and hemoglobin≥ 90 g/L;
* Liver function: Total bilirubin（TBIL）≤ 1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN for the subjects without liver metastasis; ALT and AST≤ 5×ULN for the subjects with liver metastasis;
* Kidney function: Serum creatinine ≤ 1.5 ×ULN or creatinine clearance rate ≥ 50 mL/min(Cockcroft-Gault formula);
* The subject has voluntarily signed the written informed consent form (ICF) and can comply with the study protocol;
* The female subjects of childbearing age and male subjects with fertility potential female partner agree to take reliable contraceptive measures (such as abstinence, sterilizing operation, contraceptives, injection of the contraceptive drug •medroxyprogesterone acetate or subdermal implant of contraceptives) during the study period and within 6 months after infusion of the study drugs.

Exclusion Criteria:

* Patients with brain malignant tumor, lymphoma or other malignant blood diseases;
* The subjects with symptomatic brain metastasis;
* Other malignant tumors within 5 years prior to screening (except for stage Ib or lower cervical cancer, non-invasive basal cells or squamous cell skin cancer that have been cured);
* Patients with uncontrollable ascites, pleural effusion;
* Ongoing or active systemic infection need intravenous antibiotic treatment;
* Medical history of the following diseases within 6 months before screening: myocardial infarction, unstable angina, history of coronary revascularization, congestive heart failure (New York Heart Association classification ≥ grade II), severe unstable ventricular arrhythmia, serious arrhythmia which needs drug treatment;
* The patient with hepatitis B surface antigen (HBsAg) positive and the peripheral blood HBV DNA titer ≥1× 103 copies/mL or 200 IU/ml The subject is eligible to be enrolled if HBsAg is positive and peripheral blood hepatitis B virus (HBV) DNA titer <1×103 copies/ml or 200 IU/ml and the investigator considers that the subject is at the stable stage of chronic hepatitis and the risk will not be increased for the subjects;the patient with hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody positive;
* Patients still with clinically significant electrolyte disorders that were diagnosed by the investigator before drug administration;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days for the LY01610 monotherapy (first treatment cycle of every subjects)
  The DLT of LY01610 monotherapy was obtained through the dose-increasing study of LY01610
Dose limiting toxicity (DLT) | 14 days for the LY01610 combined 5-Fu (first treatment cycle of every subjects)
  The DLT of combination of LY01610 and 5-fu was obtained through the dose-increasing study of LY01610 and 5-Fu
Maximum tolerated dose(MTD) | 21 days for the LY01610 monotherapy (first treatment cycle of every subjects)
  The MTD of LY01610 monotherapy was obtained through the single-drug dose increase study
Maximum tolerated dose(MTD) | 14 days for the LY01610 combined 5-Fu (first treatment cycle of every subjects)
  The MTD of combination of LY01610 and 5-fu was obtained through the combined dose increase study

SECONDARY OUTCOMES:
AUC | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The AUC of LY01610 monotherapy was obtained through the dose escalation and extension study，the AUC of active comparator CAMPTO® was obtained through the study，and the AUC of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
t1/2 | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The t1/2 of LY01610 monotherapy was obtained through the dose escalation and extension study，the t1/2 of active comparator CAMPTO® was obtained through the study，and the t1/2 of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
Cmax | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The Cmax of LY01610 monotherapy was obtained through the dose escalation and extension study，the Cmax of active comparator CAMPTO® was obtained through the study，and the Cmax of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
tmax | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The tmax of LY01610 monotherapy was obtained through the dose escalation and extension study，the tmax of active comparator CAMPTO® was obtained through the study，and the tmax of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
Vd | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The Vd of LY01610 monotherapy was obtained through the dose escalation and extension study，the Vd of active comparator CAMPTO® was obtained through the study，and the Vd of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
CL | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The CL of LY01610 monotherapy was obtained through the dose escalation and extension study，the CL of active comparator CAMPTO® was obtained through the study，and the CL of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
MRT | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The MRT of LY01610 monotherapy was obtained through the dose escalation and extension study，the MRT of active comparator CAMPTO® was obtained through the study，and the MRT of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
Kel | 22 days for the LY01610 monotherapy (first treatment cycle of every subjects)，5 days for the active comparator CAMPTO® (first treatment cycle of every subjects)，and 15 days for the LY01610 combined with 5-fu(first treatment cycle of every subjects)
  The Kel of LY01610 monotherapy was obtained through the dose escalation and extension study，the Kel of active comparator CAMPTO® was obtained through the study，and the Kel of LY01610 combined with 5-fu was obtained through the dose escalation and extension study.
Best Objective Response Rate | 8 weeks from enrollment
  Preliminary efficacy evaluation of LY01610 and LY01610 combined with 5-fu
Progression Free Survival | from the date of enrollment to the date of disease progression or death up to 24 months from randomisation of the subject
  Preliminary efficacy evaluation of LY01610 and LY01610 combined with 5-fu
Overall Survival | from the date of enrollment to the date of death up to 24 months from randomisation of the subject
  Preliminary efficacy evaluation of LY01610 and LY01610 combined with 5-fu

CONTACTS AND LOCATIONS:
Overall Officials: Huang jing, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Zhang B, Xu J, Wang X, Tang J, Huang J. Phase I study of liposomal irinotecan (LY01610) in patients with advanced esophageal squamous cell carcinoma. Cancer Chemother Pharmacol. 2021 Sep;88(3):403-414. doi: 10.1007/s00280-021-04294-2. Epub 2021 May 24. PMID 34031756